CLINICAL TRIAL: NCT00967837
Title: Effects of Pulsatile Intravenous Insulin Therapy on Diabetic Subjects With Non Healing Wounds
Brief Title: Effects of Pulsatile Intravenous (IV) Insulin on Wound Healing in Diabetics
Acronym: wounds
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Administrative
Sponsor: Florida Atlantic University (Other)
Collaborators: Advanced Diabetes Treatment Centers (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H09-66
Record Dates: First submitted 2009-08-06; First posted 2009-08-28 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Wound Healing; Diabetes
Keywords: Diabetes with complications; Wound healing
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin, Regular, Human; Insulin; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diabetes with non healing wounds (Experimental): To determine and monitor progress of diabetic patients with non healing wounds that have failed conventional 60 day treatment respond to pulsatile intravenous insulin therapy in improving and completing healing in non healing wounds
  Interventions: Procedure: Pulsatile Intravenous Insulin Therapy

INTERVENTIONS:
Procedure: Pulsatile Intravenous Insulin Therapy — Diabetic pts that meet trial criteria referred by an endocrinologist are given Pulsatile intravenous insulin therapy on a weekly basis. Weekly orders for insulin dosage is based upon pt response to therapy monitored by RQ and insulin resistance.
  Other Names: Humulin, Humulin R, Novolog

SUMMARY:
One of the significant complications associated with some patients with diabetes is the inability for wounds to heal regardless of enrolling and participating in a traditional wound healing program. There have been a number of anecdotal evidence presented by patients receiving pulsatile intravenous insulin therapy for other complications with non healing wounds lasting from several months to several years whose wounds healed while receiving therapy. This study was designed to specifically monitor the progress of diabetic patients who have failed traditional wound care therapy and monitor the progress of their wounds while receiving pulsatile intravenous insulin therapy.

DETAILED DESCRIPTION:
Diabetes can produce complications including the inability for wounds to heal despite participating in a traditional wound care therapy program.

At times of reduced tissue oxygen, such as when circulation is decreased, there is anecdotal evidence that pulsed IV insulin (by enabling the production of energy from glucose) may permit heart, skeletal muscle, skin, and other organs to function more normally and even to repair damage and heal. By tracking the progress in diabetic patients that have failed traditional wound care therapy who are monitored by their podiatrist or other health care professional to objectively determine the effect of pulsatile IV therapy on the rate of healing.

Independent evaluation of the wound is provided including visual examination, pictures and measurements on a weekly to bi-weekly basis.

Individuals breathe into a mask for 3-5 minutes after a rest period of 30 or more minutes. The ratio of exhaled volume of CO2 to the inhaled volume of O2 is determined as the RQ. The physiologic range is 0.7 to1.3. Individuals using fat as a primary fuel have a ratio of 0.7, protein or mixed fuels is 0.8-0.9 and carbohydrate is 0.9-1.0. Those taking excessive calories will have RQ's higher than 1.05. The RQ can be followed serially and this is done before and after each pulsatile IV insulin treatment, during the 3 successive sessions on a single treatment day. The amount of intravenous insulin and oral glucose given is determined by the RQ changes during the previous session. Pulsatile IV insulin therapy encourages the glucose metabolism in diabetics to normalize in multiple organs, especially muscle, retina, liver, kidney and nerve endings. The process fundamentally requires the administration of high dose insulin pulses similar to those found in non diabetic humans by their pancreas into the surrounding portal circulation. Oral carbohydrates are given simultaneously to augment the process and prevent hypoglycemia. The process is monitored by frequent glucose levels and respiratory quotients (RQ). RQ is measured by a metabolic cart which determines the ratio VCO2/ VO2. This ratio is specific for the fuel used at any one time by the body. The glucose levels are monitored to keep glucose levels appropriate and the RQ determines the need to readjust the infusion protocol in each patient for subsequent insulin infusion sessions.Patient is evaluated post session and discharged when stable.

Frequent monitoring of RQ is necessary as these levels change rapidly, depending on the fuel being utilized by the body. Pulsatile IV insulin therapy shifts metabolism from primarily fatty acid metabolism to primarily glucose metabolism. This shift is reflected by the increase in respiratory quotient. However during rest periods the RQ may fall back to lower levels. Therefore RQ's are done at the beginning and at the end of each insulin infusion session of 1 hour in order to appropriately monitor and adjust insulin and carbohydrate loads to reach optimal activation in each session

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with type 1 or type 2 diabetes
* taking oral and/or insulin for diabetes control
* endocrinologist must assess and approve pt for participation in study
* ability to swallow without difficulty
* ability to meet weekly time and testing requirements for this study

Exclusion Criteria:

* inability to do testing required for study including regular scheduled visits for independent review of non healing wound including assessment, pictures and measurements
* lack of intravenous access
* alcohol abuse, drug addiction or the use of illegal drugs
* positive HIV
* active liver disease
* in active treatment for cancer including radiation or chemotherapy
* inability to breathe into machine for respiratory quotients to monitor progress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2006-01; Primary Completion 2012-01 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To measure progress of wound healing in subjects that have failed conventional wound care healing treatments for 60 days | Monitoring of wound is done at baseline and weekly follow up visits including visual examination, pictures of wound and measurements

CONTACTS AND LOCATIONS:
Overall Officials: Betty Tuller, PhD, Principal Investigator — Florida Atlantic University
Locations (1):
- Florida Atlantic University, Boca Raton, Florida, United States